CLINICAL TRIAL: NCT07017543
Title: Patient Capacity and Dynamic Aspects of the Psychotherapeutic Process Impacting the Course and Outcomes of Treatment
Brief Title: Dynamics of Psychotherapy and Treatment Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital in Krakow (Other)
Responsible Party: Principal Investigator, Benita Wielgus, MSc, University Hospital in Krakow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1072.6120.189.2022
Record Dates: First submitted 2025-04-28; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Mental Disorders; Neurotic Disorders; Personality Disorders
Keywords: therapeutic alliance; insight; resilience; group therapy; neurotic symptoms; treatment oucome; changes in treatment; mindfulness; process-outcome research
MeSH Terms: conditions — Mental Disorders; Neurotic Disorders; Personality Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trait-like and state-like components of therapeutic alliance and insight influencing psychotherapy o (Other): Patients diagnosed with neurotic and personality disorders were assessed at the 1st, 4th, 8th, and 12th week of treatment using the psychological assessment measures.
  Interventions: Other: Psychotherapy Process-Outcome Study in Group Therapy

INTERVENTIONS:
Other: Psychotherapy Process-Outcome Study in Group Therapy — A manualized group dynamic psychotherapy conducted at the University Hospital in Kraków, focused on monitoring and enhancing therapeutic alliance and insight development. The intervention targeted patients diagnosed with neurotic and personality disorders. Psychological assessments were conducted at weeks 1, 4, 8, and 12 to track changes in symptoms, resilience, alliance, and insight. The psychotherapy emphasized the interplay between trait-like and state-like components of alliance and insight and their relationship to therapeutic outcomes (symptom reduction and resilience enhancement).
  Other Names: Group Psychotherapy Focused on Therapeutic Alliance and Insight; Alliance-Focused Group Therapy; Insight-Oriented Group Therapy; Psychodynamic Group Therapy Monitoring Alliance and Insight Development; Resilience-Focused Group Dynamic Psychotherapy

SUMMARY:
The study is a 3-month controlled trial that aims to measure changes in patient's capacity (mindfulness, resilience, insight, working alliance) and intensity of neurotic symptoms. The following tools are used: the Freiburg Mindfulness Inventory, the Psychological Insight Questionnaire, the Connor-Davidson Resilience Scale - Short Version, the Working Alliance Inventory - Short Version and the "O" Symptom Questionnaire. During 12-week group intervention patients are asked to fill in the appropriate set of questionnaires four times (at the beginning, two times between and at the end of treatment). The study is conducted in the Psychotherapy Unit of University Hospital in Krakow.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic criteria for neurotic disorders (ICD-10: F40-F48.9) or personality disorders of mild to moderate severity (ICD-10: F60-F61)
* obtaining informed consent for participation in the study
* being over the age of 18

Exclusion Criteria:

* diagnosis of psychotic and/or organic disorders as well as active addictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resilience Level Assessed by the Connor-Davidson Resilience Scale Short Version (CD-RISC-10) | Week 1 (pre-treatment); Week 4 (1 month of treatment); Week 8 (2 months of treatment); Week 12 (post-treatment; end of 3-month therapy cycle)
  Connor-Davidson Resilience Scale Short Version (CD-RISC-10) is a 10-item scale used to assess resilience, defined as the ability to cope with stress in response to challenging experiences. The full CD-RISC consists of 25 items and has a five-factor structure, both versions displaying sound psychometric properties. Observations made during the development of the original scale indicate that resilience can be modified and improved through appropriate interventions, and greater improvement in resilience scores corresponds to more significant overall treatment outcomes. CD-RISC is one of the most frequently used tools to measure resilience. This study employed the short version, CD-RISC-10, which includes two factors labeled as Endurance and Perseverance. The CD-RISC-10 uses a 5-point Likert scale to assess resilience.
Neurotic Symptoms Questionnaire "O" (SQ-O) | Week 1 (pre-treatment); Week 4 (1 month of treatment); Week 8 (2 months of treatment); Week 12 (post-treatment; end of 3-month therapy cycle)
  The Symptoms Questionnaire "O" (SQ-O), a validated 187-item self-report tool used to measure the severity of neurotic symptoms across affective, somatic, and behavioral domains. The checklist includes 14 subscales covering different areas of neurotic psychopathology. The SQ-O can be used both diagnostically, to assess the overall severity of symptoms (cut-off scores are sex-adjusted; scores above 165 for men and 200 for women indicate symptoms exceeding the norm), as well as a measure of treatment-related change. This study focused on the overall scale scores measured at specified time points, without analyzing changes in individual subscales. Each item is scored dichotomously (0 = no, 1 = yes).
Psychological Insight Assessed by the Psychological Insight Questionnaire (PIQ) | Week 1 (pre-treatment); Week 4 (1 month of treatment); Week 8 (2 months of treatment); Week 12 (post-treatment; end of 3-month therapy cycle)
  Psychological Insight Questionnaire (PIQ) is a tool used to assess insight, defined as a series of realizations and discoveries related to personality, relationships, behavioral patterns, and emotions. The questionnaire consists of 23 items rated on a 6-point Likert scale (from 0 - none/not at all to 5 - extreme) to indicate the intensity of each experienced state over the last 7 days. The scale includes two subscales: (1) Avoidance and Maladaptive Patterns Insights and (2) Goals and Adaptive Patterns Insights, both of which demonstrate satisfactory internal consistency (Cronbach's α = 0.93 and 0.85, respectively). Although initially developed to explore the acute and lasting effects of psychedelic use, the content, sound psychometric properties, and simplicity of the PIQ encourage its use in other areas where psychological insight may be critical in predicting psychotherapy outcomes.
Therapeutic Alliance Level Assessed by the Working Alliance Inventory - Short Revised (WAI-SR) | Week 1 (pre-treatment); Week 4 (1 month of treatment); Week 8 (2 months of treatment); Week 12 (post-treatment; end of 3-month therapy cycle)
  Working Alliance Inventory - Short Revised (WAI-SR) is a 12-item revised measure assessing the quality of the therapeutic alliance as perceived by the patient. Extensive research has confirmed its effectiveness in predicting treatment outcomes. Most researchers recommend using the overall score, as the two identified subscales - Goal/Task and Bond - strongly correlate, which could interfere with accurate interpretation. The WAI-SR uses a 5-point Likert scale to assess the strength of the therapeutic alliance.
Freiburg Mindfulness Inventory - Short Form (FIU-14) | Week 1 (pre-treatment); Week 4 (1 month of treatment); Week 8 (2 months of treatment); Week 12 (post-treatment; end of 3-month therapy cycle)
  The Freiburg Mindfulness Inventory - Short Form (FIU-14) is a 14-item self-report scale designed to measure mindfulness as a general psychological trait. Mindfulness is described as a personal trait of being mindful of the moment-by-moment experience. Some of the features of mindfulness include openness, receptiveness, curiosity, and a nonjudgmental attitude. It assumes that an open and attentive individual is more in touch with feelings and experiences. Fourteen items of the questionnaire define mindfulness as a process of regulating attention. The items are rated on a 4-point Likert scale, from 1 = "rarely" to 4 = "almost always". The reliability measure of this short version is acceptable (Cronbach's alpha between 0.79 and 0.86).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Krakow, Małopolska, Poland

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07017543/Prot_SAP_ICF_000.pdf